CLINICAL TRIAL: NCT06793826
Title: Post-marketing Surveillance Study for the Safety of Hexaxim®, a DTaP-IPV- HB-PRP~T Vaccine Administered to Infants From 2 Months of Age in Republic of Korea
Brief Title: Post-marketing Surveillance Study for the Safety of a DTaP-IPV- HB-PRP~T Vaccine in Republic of Korea
Status: Recruiting | Type: Observational
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: A3L46; U1111-1266-4935 (Registry Identifier: ICTRP)
Record Dates: First submitted 2025-01-21; First posted 2025-01-27 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Hepatitis B; Haemophilus Influenzae Type b Immunisation
MeSH Terms: conditions — Hepatitis B | interventions — DTaP-IPV-HB-PRP-T vaccine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — max 1000 characters
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort: Infants from 2 months of age vaccinated with 1 dose of Hexaxim on the day of enrollment
  Interventions: Biological: DTaP-IPV-Hep B-PRP-T combined vaccine

INTERVENTIONS:
Biological: DTaP-IPV-Hep B-PRP-T combined vaccine — prefilled syringe injection intramuscular
  Other Names: Hexaxim®

SUMMARY:
Primary objectives:

To investigate the incidence of adverse events occurred following administration of Hexaxim in infants from 2 months of age under routine clinical practice, as per approved indications

DETAILED DESCRIPTION:
The duration of each enrolled participant's participation in the study will be up to 36 or 43 days.

ELIGIBILITY:
Inclusion Criteria:

* An infant aged 2 months or more on the day of enrollment
* Infant whose parent or legal representative has signed and dated the ICF
* Receipt of 1 dose of Hexaxim on the day of enrollment according to the approved local product label (regardless of vaccinated dose)

Exclusion Criteria:

* Deviational use (off-label vaccination) from the approval local product label of Hexaxim
* Previous history of enrollment in this study
* Participation at the time of study enrollment (or in the 4 weeks preceding the enrollment) or planned participation during the present study period in a clinical study investigating a vaccine, drug, medical device or medical procedure

Ages: 2 Months to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants aged 2 months or more will be recruited after vaccination with Hexaxim as per a routine healthcare visit and according to approved local product labeling, at study centers (general hospitals or clinics located in Korea). The number of subjects to enroll per site (10 sites) will be defined with each investigator
Sampling Method: Non-Probability Sample
Enrollment: 690 (Estimated)
Dates: Start 2025-01-17 (Actual); Primary Completion 2026-04-13 (Estimated); Study Completion 2026-04-13 (Estimated)

PRIMARY OUTCOMES:
Number of participants reporting immediate adverse events/adverse drug reactions (AEs/ADRs) | Within 30 minutes post-vaccination
  Unsolicited (spontaneously reported) systemic AEs/ADRs
Number of participants reporting serious adverse events / adverse drug reactions (SAEs / SADRs) | Up to 43 days post-vaccination
  SAEs and SADRs
Number of participants reporting solicited injection site and systemic reactions | Up to 7 days post-vaccination
  Solicited injection site reactions: tenderness; erythema; site swelling Solicited systemic reactions: vomiting; crying abnormal; drowsiness; appetite loss; irritability
Number of participants reporting unsolicited non-serious AEs/ADRs | Up to 28 days post-vaccination
  Unsolicited non-serious AEs and ADRs

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (2):
- South Korea (2):
  - Investigational Site Number : 002, Cheonan
  - Investigational Site Number : 001, Seoul

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org